CLINICAL TRIAL: NCT00536809
Title: A Phase I/II Study of Lapatinib in Combination With Oxaliplatin and Capecitabine in Subjects With Advanced or Metastatic Colorectal Cancer
Brief Title: Phase I/II Study of Lapatinib in Combination With Oxaliplatin and Capecitabine in Subjects With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGF108991
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms, Colorectal
Keywords: Metastatic Colorectal Cancer; oxaliplatin; fluoropyrimidines cancers; Advanced Colorectal Cancer; capecitabine; lapatinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lapatinib; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I (Experimental): Dose escalation of lapatinib along with capecitabine and oxaliplatin until the maximum tolerated dose is reached.
  Interventions: Drug: oxaliplatin
- Phase II (Experimental): Treatinng subjects at the maximum tolerated dose of lapatinib, capecitabine, and oxaliplatin
  Interventions: Drug: lapatinib; Drug: oxaliplatin; Drug: capecitabine

INTERVENTIONS:
Drug: lapatinib — onced daily Days 1-21
  Arms: Phase II
Drug: oxaliplatin — Day one of each cycle
Drug: capecitabine — given BID days 1-14
  Other Names: lapatinib; oxaliplatin
  Arms: Phase II

SUMMARY:
The purpose of this study is to determine the highest, tolerated dose level and safety of lapatinib, capecitabine and oxaliplatin in subjects with advanced cancer and to determine the clinical activity of the combination of drugs in subjects with previously untreated advanced or metastatic colorectal cancer.

ELIGIBILITY:
Inclusion criteria

1. 18 years of age or older.
2. A female is eligible to enter and participate in the study if she is of:

   * Non-child-bearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:
   * Has had a hysterectomy, or
   * Has had a bilateral oophorectomy (ovariectomy), or
   * Has had a bilateral tubal ligation, or
   * Is considered post-menopausal (defined as amenorrheic for greater than or equal to 1 year).
   * Childbearing potential, has a negative serum pregnancy test at Screening and agrees to one of the following from 2 weeks prior to enrolment and continue through the post-study visit:
   * Complete abstinence from sexual intercourse
   * Oral Contraceptive, either combined or progestogen alone (must use a back up method, if have taken for less than 3 cycles)
   * Injectable progestogen
   * Implants of levonorgestrel
   * Estrogenic vaginal ring
   * Percutaneous contraceptive patches
   * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
   * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
   * Double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository)
3. Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2.
4. Provided written informed consent.
5. Hemoglobin greater than or equal to 8 gm/dL (5 nmol/L), if clinically stable.
6. Absolute neutrophil count greater than or equal to 1,500/mm^3 (1.5 x 109/L).
7. Calculated creatinine clearance (CrCl) greater than or equal to 50 mls/min.
8. Total bilirubin less than or equal to 1.25 times the institutional upper limit of normal (ULN).
9. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2 times the ULN. For subjects with liver metastases: AST or ALT less than or equal to 5 times the ULN.
10. LVEF greater than or equal to 50% or greater than or equal to LLN for the institution based on multiple gated acquisition scan (MUGA) or echocardiogram (ECHO).

    Specific to Phase I:
11. Recurrent, advanced, or metastatic cancer that is known to be potentially responsive to treatment with fluoropyrimidines or oxaliplatin. Examples include gastrointestinal tumors, HER2 (ErbB2)-positive breast cancer, and lung cancers.
12. Received less than or equal to 3 prior chemotherapy regimens without pelvic radiotherapy or less than or equal to 2 prior chemotherapy regimens if received pelvic radiotherapy.
13. Platelet count greater than or equal to 75,000/mm^3 (75 x 109/L).

    Specific to Phase II:
14. Histologically-confirmed, measurable advanced or metastatic CRC previously untreated in the metastatic setting or more than 6 months post an oxaliplatin-containing adjuvant therapy.
15. Archived paraffin-embedded tumor tissue must be available for biomarker analysis.
16. Platelet count greater than or equal to 100,000/mm^3 (100 x 109/L).

Exclusion Critera:

1. Pregnant or lactating female.
2. Prior resection of the small bowel.
3. Brain metastases that require additional treatment.
4. Medically unfit for the study as a result of the medical interview, physical exam, or screening investigations.
5. Taking any medication on the prohibited medications list (see Section 9.2).
6. History of drug or other allergy, which, in the opinion of the Investigator, contraindicates participation.
7. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs. These include other anilinoquinazolines, such as gefitinib [Iressa], or erlotinib [Tarceva]. The subject has received treatment with any investigational drug in the previous four weeks.
8. Treatment with any biologic, cytotoxic, radiation , or hormonal (other than for contraception or replacement) therapy within four weeks. Treatment with hormones with short half-lives is allowed up to 1 week prior to study treatment after consultation with GSK medical monitor.
9. Major surgery within the previous two weeks unless in the opinion of the Investigator, the subject has recovered sufficiently to begin study treatment.
10. Physiological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
11. Receiving concurrent coumadin therapy. Minidose coumadin for maintenance of catheters (0.5 to 1.0 mg/day), and other anticoagulation therapy are allowed on study. Subjects receiving minidose coumadin must have prothrombin time (PT) or International normalized ratio (INR) and partial thromboplastin time (PTT) within 1.2 times the ULN.
12. History of uncontrolled or symptomatic angina, arrhythmias, or congestive heart failure.
13. Corrected QT interval (QTc) greater than 450 msecs.

    Specific to Phase I:
14. Residual chemotherapy related toxicity of greater than or equal to Grade 2 that is clinically felt likely to be exacerbated by the treatment regimen.

    Specific to Phase II (amendment written after the completion of Phase 1):
15. Have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-09-26 (Actual); Primary Completion 2008-10-31 (Actual); Study Completion 2008-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Dennie TW, Fleming RA, Bowen CJ, Dar MM, Alberti D, Oliver K, Loconte N, Mulkerin D, Holen KD. A phase I study of capecitabine, oxaliplatin, and lapatinib in metastatic or advanced solid tumors. Clin Colorectal Cancer. 2011 Mar 1;10(1):57-62. doi: 10.3816/CCC.2011.n.008. PMID 21609937
- See also: Results for study EGF108991 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/EGF108991?search=study&search_terms=108991#rs

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase I/II study. Enrollment of Phase I was complete; however, Phase II of the study was terminated early due to lake of interest by sites in participating. Only 2 of the 15 planned participants were enrolled prior to termination.
Groups:
- Lapatinib/Oxaliplatin/Capecitabine: Phase I: Dose escalation to a maximum tolerated dose of lapatinib 1000 milligrams (mg)/day administered orally on Days 1-21, oxaliplatin 130 mg/square meters (m^2) administered intravenously on Day 1, and capecitabine 1500 mg/m^2/day on Days 1-14 of a 21-day cycle. Phase II: Lapatinib 1000 mg/day administered orally on Days 1-21, oxaliplatin 130 mg/m^2 administered intravenously on Day 1, and capecitabine 1500 mg/m^2/day on Days 1-14 of a 21-day cycle.
Period: Phase I (Dose-finding Phase)
Arm/Group | Lapatinib/Oxaliplatin/Capecitabine
Started | 10
Completed | 10
Not Completed | 0
Period: Phase II
Arm/Group | Lapatinib/Oxaliplatin/Capecitabine
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Referred for surgical resection | 1

BASELINE CHARACTERISTICS:
Groups:
- Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2: Lapatinib (Lap.) 1000 milligrams (mg)/day administered orally on Days 1-21, oxaliplatin 130 mg/square meters (m^2) administered intravenously on Day 1, and capecitabine 1500 mg/m^2/day on Days 1-14 of a 21-day cycle
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] — Baseline participants include the 10 participants who completed Phase I, and the 2 who were enrolled into Phase II before the study was terminated.
  years | 59.9 [36 to 78]
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline participants include the 10 participants who completed Phase I, and the 2 who were enrolled into Phase II before the study was terminated.
  Participants
    Female | 11
    Male | 1
Race/Ethnicity, Customized [Number; unit: participants] — Baseline participants include the 10 participants who completed Phase I, and the 2 who were enrolled into Phase II before the study was terminated.
  participants
    White/Caucasian/European heritage | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response in Phase II
Description: The overall response is defined as the number of participants whose tumor response was classified as a complete response (CR; disappearance of all target lesions) or partial response (PR; 30% decrease in the sum of the longest diameter of target lesions) per Response Evaluation Criteria in Solid Tumors. Response was measured for participants in Phase II only. To determine response, radiographic images were taken at baseline, 8 weeks, and every 8 weeks thereafter until the participant withdrew from the study.
Time Frame: Baseline to response (up to 135 days)
Population: All-Treated Population for Phase II: all participants who received at least one dose of lapatinib
Measure: Number; unit: participants
Groups:
- Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2: Lapatinib (Lap.) 1000 milligrams (mg)/day administered orally on Days 1-21, oxaliplatin 130 mg/square meters (m^2) administered intravenously on Day 1, and capecitabine 1500 mg/m^2 administered orally twice a day on Days 1-14 of a 21-day cycle
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 2
participants | 2

2. Secondary Outcome: Relationship Between Pretreatment Plasma TS mRNA and Pretreatment Tumor TS mRNA in Colon Tumor Biopsies.
Description: Exploring if there is an association with a reduction in thymidylate synthase (TS) gene expression in both plasma and tumor prior to treatment and increased sensitivity in clinical activity. This analysis was not completed due to the study being closed early and the small number of participants enrolled in Phase II.
Time Frame: Plasma TS mRNA is collected at screening. Pre-treatment tumor sample can be archived tissue if collected within 5 years from screening; if not, tumor sample should be collected at screening.
Population: All-Treated population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

3. Secondary Outcome: Effect of Lapatinib, Oxaliplatin, and Capecitabine on Plasma TS mRNA and the Relationship Between Plasma TS mRNA and Clinical Response
Description: A possible association between a reduction in thymidylate synthase (TS) gene expression and increased sensitivity in clinical activity was to be explored. This analysis was not completed due to the study being closed early and the small number of participants enrolled in Phase II.
Time Frame: Blood samples were collected to determine TS levels at screening phase; Days 43 and 85; after every 2 cycles of treatment (+/- 3 days); and at discontinuation (if possible).
Population: All-Treated population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

4. Secondary Outcome: Tumor-derived Biomarkers (Encoded in Protein or RNA) Associated With Clinical Outcome to Treatment
Description: Exploring tumor-derived biomarkers including TS, DPD, TP, EGFR (ErbB1), and additional downstream markers involved in the mechanism of action of each compound (e.g., ERCC1) and comparison to clinical response. This analysis was not completed due to the study being closed early and the small number of participants enrolled in Phase II.
Time Frame: Pre-treatment tumor sample should have been provided for the most recent biopsy (not older than 5 years) prior to dosing. The post-treatment sample is suggested, not mandatory, and should have been collected at 43 +/-3 days.
Population: All-Treated population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

5. Secondary Outcome: Genetic Aberrations in Somatic (Tumor) DNA Derived From the Tumor Tissue Biopsies That May Associate With Clinical Outcomes in Response to Therapy
Description: DNA sequencing was done to identify genetic aberrations in somatic (tumor) DNA that may associate with clinical outcomes in response to therapy. This analysis was not completed due to the study being closed early and the small number of participants enrolled in Phase II.
Time Frame: Pre-treatment tumor sample should have been provided for the most recent biopsy (not older than 5 years) prior to dosing. The post-treatment sample is suggested, not mandatory, and should have been collected at end of Cycle 2, +/-3 days from Cycle 3.
Population: All-Treated population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

6. Secondary Outcome: Genetic Variants in Germline (Host) DNA and Comparison to the Efficacy and Safety of the Study Drugs
Description: This outcome measure was conducted to investigate a possible genetic relationship to handling or response to lapatinib, oxaliplatin, and capecitabine. This measure was not analyzed due to the small number of participants who signed the optional pharmacogenetics consent.
Time Frame: Optional pharmacogenetics sample may be collected at any time during the study after consent has been obtained; however, it is recommended that it be collected at the earliest time point possible
Population: Participants in the All-Treated Population who signed a PGx informed consent.
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

7. Secondary Outcome: Progression-free Survival (PFS) After Lapatinib, Oxaliplatin, and Capecitabine Administered at the MTD Level of Phase II
Description: Both participants that entered Phase II of the study were censored for progression-free survival. Progression-free survival (PFS) is defined as the time from first dose until the first documented sign of disease progression or death due to any cause. For participants who do not progress or die, PFS was censored at the time of last radiological scan preceding the initiation of alternative anti-cancer therapy. Of the 2 participants in Phase II of the study, one discontinued due to adverse events, and the other was referred for a surgical resection.
Time Frame: Date of the first dose of study drug to the date of documented and confirmed progression by clinical, radiographic, or biochemical criteria, whichever occurred earliest, or to date of death due to any causes (up to 135 Days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline to Study Completion in Weight
Description: Each on-study and follow-up laboratory parameter and vital sign was compared to the participant's baseline values to investigate what changes occurred. This analysis was not completed due to the study being closed early and the small number of participants enrolled in Phase II.
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline to Study Completion in Heart Rate
Description: as for outcome 8
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline to Study Completion in Blood Pressure
Description: as for outcome 8
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline to Study Completion in Hemoglobin and Neutrophils
Description: as for outcome 8
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

12. Secondary Outcome: Change From Baseline to Study Completion in White Blood Cells and Platelets
Description: as for outcome 8
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline to Study Completion in Prothrombin Time and Partial Thromboplastin Time
Description: as for outcome 8
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

14. Secondary Outcome: Change From Baseline to Study Completion in International Normalized Ratio
Description: as for outcome 8
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

15. Secondary Outcome: Change From Baseline to Study Completion in Sodium, Potassium, and Calcium
Description: as for outcome 8
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

16. Secondary Outcome: Change From Baseline to Study Completion in Creatinine, Total Bilirubin, and Direct Bilirubin
Description: as for outcome 8
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

17. Secondary Outcome: Change From Baseline to Study Completion in Creatinine Clearance
Description: as for outcome 8
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

18. Secondary Outcome: Change From Baseline to Study Completion in Aspartate Aminotransferase, Alanine Aminotranferease, and Alkaline Phosphatase
Description: as for outcome 8
Time Frame: Baseline to study completion (up to 135 days)
Population: All-Treated Population for Phase II
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Phases I and II
Description: GSK typically summarizes all AEs and all SAEs. The SAE summary will include participants with only an SAE. The data summarized below under the heading Other AEs (non-serious) are actually a summary of all AEs, which does include some SAEs.
Arm/Group | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2 (N=12)
Hypokalemia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 1
Dizziness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lap. 1000 mg/Oxaliplatin 130 mg/m^2/Capecitabine 1500 mg/m^2 (N=12)
Diarrhoea (Gastrointestinal disorders) | 12
Anorexia (Metabolism and nutrition disorders) | 10
Nausea (Gastrointestinal disorders) | 10
Peripheral sensory neuropathy (Nervous system disorders) | 9
Vomiting (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 8
Dizziness (Nervous system disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 4
Weight decreased (Investigations) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Anxiety (Psychiatric disorders) | 2
Blood albumin decreased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Hyperbilirubunaemia (Hepatobiliary disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Asthenia (General disorders) | 1
Blindness transient (Eye disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Depression (Psychiatric disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Eye pain (Eye disorders) | 1
Headache (Nervous system disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Injection site reaction (General disorders) | 1
Insomnia (Psychiatric disorders) | 1
Laryngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Left ventricular dysfunctionation (Cardiac disorders) | 1
Mucosal inflammation (General disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Oedema (General disorders) | 1
Oesophageal pain (Gastrointestinal disorders) | 1
Oral candidiasis (Infections and infestations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pyrexia (General disorders) | 1
Somnolence (Nervous system disorders) | 1
Thrombosis (Vascular disorders) | 1
Ventricular tachycardia (Vascular disorders) | 1
Vision blurred (Eye disorders) | 1
Weight increased (Investigations) | 1
Hyperaesthia (Nervous system disorders) | 1
Hyporcalceamia (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
Phase II of the study was terminated due to lake of interest. Two participants were enrolled prior to termination. Due to the small sample size in Phase II, the data were not analyzed. The two participants' data were analyzed with Phase I data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.